CLINICAL TRIAL: NCT04590196
Title: Effect of Oral Curcumin Supplementation on Choriocapillaris and Drusen Characteristics Measured by Multimodal Retinal Imaging in Dry Age-related Macular Degeneration (AMD) Patients
Brief Title: Effect of Oral Curcumin Supplementation in Dry Age-related Macular Degeneration (AMD) Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: VitreoRetinal Surgery Foundation (Unknown); Illinois Society for the Prevention of Blindness (Unknown)
Responsible Party: Principal Investigator, Jennifer I. Lim, Physician Ophthalmology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-0566; 096625 (Other Grant/Funding Number: Illinois Society for the Prevention of Blindness); 098928 (Other Grant/Funding Number: VitreoRetinal Surgery Foundation)
Record Dates: First submitted 2020-10-04; First posted 2020-10-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment (Experimental)
  Interventions: Drug: Longvida curcumin
- control (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Longvida curcumin — longvida curcumin verdure sciences formulation
  Arms: treatment
Other: placebo — Composition of Placebo :
  95.66% Maltodextrin 0.34% Sunset Yellow Color 0.06% Tartrazine Food Color 3.91% Silicon Dioxide
  Arms: control

SUMMARY:
Nutrition plays an important role in preventing progression of dry age related macular degeneration (AMD), a disease of aging that leads to drusen deposits in the macula causing significant decrease in vision. Drusen contains amyloid protein which is inhibited by curcumin, a natural plant based antioxidant. Oral Longvida curcumin has been shown to accumulate in the retina of human subjects within 10 days of supplementation. This study aims to investigate the duration of oral curcumin supplementation needed to see clinical impact in reducing volume and number of drusen and decreasing choriocapillaris density loss or flow impairment in dry AMD patients. Patients will be given a 12-month course of oral Longvida curcumin and clinical impact will be measured by multimodal retinal imaging (fundus photos, OCT and OCT-A) at day 0, month 3, month 6, and month 12 of supplementation. Previous small studies have shown change in drusen size within 4 6months of curcumin supplementation, given that drusen can naturally fluctuate in size, we want to have a longer study period with a control group to better understand the effects of curcumin on drusen characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years old BCVA 20/20 to 20/400 Dry AMD with many large (>300 μm in diameter and more than 100 μm in height) soft drusenoid PEDs

Exclusion Criteria:

* presence (or history) of significant geographic atrophy or choroidal neovascularization in either eye; history of eye surgery (other than cataract extraction) within 90 days, history of BRVO/CRVO, Macular hole, pathologic myopia, uveitis, pseudovitelliform maculopathy will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Drusen volume | baseline, 3month, 6month, 12 month timepoints
  Quantify change in volume of drusen/drusenoid pigment epithelial detachments at day 0, month 3, month 6, month 12 by comparing fundus photos and OCT images obtained at these time points

SECONDARY OUTCOMES:
Drusen size | baseline, 3month, 6month, 12 month timepoints
  Quantify change in size of drusen/drusenoid pigment epithelial detachments at day 0, month 3, month 6, month 12 by comparing diameter of drusen in OCT images obtained at these time points

CONTACTS AND LOCATIONS:
Overall Officials: Yekaterina Joltikov, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Illinois eye and ear infirmary, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No